CLINICAL TRIAL: NCT02489864
Title: The Effect of Terlipressin in the Prevention of Type 2 Hepatorenal Syndrome by Improving Mean Arterial Pressure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chan Xie, Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005004
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Hepatorenal Syndrome
Keywords: Terlipressin; mean arterial pressure; type 2 HRS
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Terlipressin

ARMS (2):
- Terlipressin and albumin (Active Comparator): Patients in this group received terlipressin as an intravenous bolus of 0.5 mg every 6 h. If a significant reduction in serum creatinine level (≥1 mg/dL) was not observed during 3-day period, the dose of terlipressin was increased in a stepwise fashion every 3 days to a maximum of 2 mg every 6 hour.
  albumin (Albumin 20 percent; Instituto Grífols, Barcelona, Spain) was given at a dose of 10 gram per day.
  Interventions: Drug: Terlipressin
- Albumin (Placebo Comparator): Only albumin (Albumin 20 percent; Instituto Grífols, Barcelona, Spain) was given at a dose of 10 gram per day.
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin

SUMMARY:
Appreciation of the central role for arterial vasodilatation in the pathogenesis of hepatorenal syndrome (HRS) has led to routine use of vasoconstrictors in combination with albumin as a medical therapy for HRS. Terlipressin have been explored but the optimal approach for such therapies has not yet been established. As compared with albumin, treatment with terlipressin and albumin is effective in improving renal function in patients with cirrhosis and hepatorenal syndrome. Our previous study showed that mean arterial pressure (MAP) is a predictor of hepatorenal syndrome occurrence in cirrhotic patients with ascites. The purpose of this study was to examine the role of targeting an early and substantial increase in mean arterial pressure in the prevention of type 2 HRS.

ELIGIBILITY:
Inclusion Criteria:

1. cirrhosis as diagnosedby liver biopsy or clinical, biochemical, ultrasound,and/or endoscopic findings;
2. type 2 HRS with a MAP decrees for at least 10mmHg compared to basal blood pressure ;
3. age 18 to65 years;
4. absence of severe bacterial infection associated with findings of systemic inflammatory response as diagnosedby the presence of at least 2 of the following criteria: body temperature <36°C or >38°C, heart rate >90 beats/min, respiration rate>20/min, and white-cell count <4 or >12 X106/L or >6% of band forms; patients with bacterial infections, however, could be included in the study if renal failure persisted after infection resolution;
5. the absence of cardiovascular diseases and any extra hepatic disease that could affect the short-term prognosis;
6. the absence of findings suggestive of organic nephropathy;
7. the absence of advanced hepatocellularcarcinoma.

Exclusion Criteria:

1. Patients with history of coronary artery disease
2. Cardiomyopathy
3. Ventricular arrhythmia
4. Obstructive arterial disease of limbs -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
HRS incidence rate | one year

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China